CLINICAL TRIAL: NCT04730037
Title: An Investigator-initiated, Multicenter, Phase 3, Randomized, Single-blind, Double-dummy, Parallel-group Study of Evaluate the Efficacy and Safety of Edoxaban Versus Warfarin (Vitamin K Antagonist) in Subjects With Chronic Thromboembolic Pulmonary Hypertension Taking Warfarin (Vitamin K Antagonist) at Baseline: KABUKI
Brief Title: Clinical Trial to Investigate Safety and Efficacy of Edoxaban in Patients With CTEPH (KABUKI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyushu University (Other)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kohtaro Abe, Department of Cardiovascular Medicine, Faculty of Medical Sciences, Kyushu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTR225-01
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: CTEPH
Keywords: Edoxaban; DOAC; Wafrarin; Anticoagulation
MeSH Terms: interventions — edoxaban; Warfarin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edoxaban group (Active Comparator)
  Interventions: Drug: Edoxaban; Drug: Warfarin Potassium placebo
- Warfarin group (Active Comparator)
  Interventions: Drug: Warfarin Potassium; Drug: Edoxaban placebo

INTERVENTIONS:
Drug: Edoxaban — - Edoxaban 30 mg/60 mg tablet according to body weight. 60 kg or less: 30 mg once daily, over 60 kg: 60 mg once daily, reduced to 30 mg once daily depending on renal function and concomitant medications
  Arms: Edoxaban group
Drug: Warfarin Potassium — - Warfarin K 1 mg tablets once daily (Dose adjusted with target PT-INR of 1.5-2.5)
  Arms: Warfarin group
Drug: Warfarin Potassium placebo — - Warfarin K 1 mg placebo tablets once daily
  Arms: Edoxaban group
Drug: Edoxaban placebo — - Edoxaban 30 mg/60 mg placebo tablet according to body weight. 60 kg or less: 30 mg once daily, over 60 kg: 60 mg once daily, reduced to 30 mg once daily depending on renal function and concomitant medications
  Arms: Warfarin group

SUMMARY:
This is phase III trial to evaluate whether edoxaban, a direct factor Xa inhibitor, is noninferior to warfarin in preventing worsening of chronic thromboembolic pulmonary hypertension (CTEPH).

ELIGIBILITY:
Inclusion Criteria:

1. Patient who once* diagnosed with CTEPH based on at least 2 imaging study (VQ scan, CT pulmonary angiogram, or catheter-based pulmonary angiogram) and hemodynamic criteria (MPAP >=25 mmHg and PAWP =< 15 mmHg). *Patients treated with PEA, BPA, or vasodilators, who do not meet hemodynamic criteria at the registration, are eligible.
2. Patients who are not planned to require increased / changed / discontinuation of PEA, BPA, or pulmonary vasodilators within 12months
3. Stable administration of vitamin K antagonists
4. WHO functional class I-III
5. Patients who meet A) B)and C) by 90 days prior to baseline. A)No addition, reduction, or change of endothelin antagonists, soluble guanylate cyclase stimulants, phosphodiesterase-5 inhibitors, prostacyclin, and its derivatives, or calcium antagonists. B)Appropriate anticoagulants have been continued. C)No BPA has been done.
6. Patients who have not undergone PEA from 180 days prior to baseline right heart catheterization to the start date of study drug administration
7. Patients with a 6-minute walking distance >=150m

Exclusion Criteria:

1. Patients with severe lung disease (FEV1.0/FVC < 60% or %TLC < 60%)
2. Patients with acute or chronic disabilities that interfere with clinical trial requirements
3. Patients with acute symptomatic PE within 180 days prior to the start of study drug administration
4. Patients with congenital heart disease who have not undergone radical surgery
5. Patients who cannot provide informed consent due to mental disorders, dementia, or other illnesses
6. Patients with advanced cancer
7. Patients with a life expectancy of less than 1 year
8. Patients with active hemorrhagic lesions
9. Patients with comorbidities requiring vitamin K antagonist
10. Patients receiving other study drug within 30 days prior to randomization
11. Patients with renal dysfunction (Ccr 15 mL/min)
12. Patients with liver dysfunction (Child-Pugh B or C)
13. Females of reproductive age not using an acceptable form of contraception/Pregnant/Breastfeeding
14. Patients contraindicated for edoxaban or warfarin
15. Patients with hypersensitivity to any of the drug

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Ratio of 1-year resting PVR to baseline resting PVR | Week 48 of treatment

SECONDARY OUTCOMES:
Percentage of cases with worsening of CTEPH | Throughout the study duration(up to week48)
Change from baseline in 6-minute walk distance | Week16, 32, 48 of treatment
Change from baseline in WHO functional class | Week16, 32, 48 of treatment
Change from baseline in NT-proBNP | Week16, 32, 48 of treatment
Percentage of cases with clinically relavant bleeding (ISTH 2015 definition) | Throughout the study duration(up to week48)

CONTACTS AND LOCATIONS:
Overall Officials: Kohtaro Abe, Principal Investigator — Kyushu University Hospital
Locations (1):
- Kyushu University Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No
Data are available upon reasonable request. The deidentified participant data collected in this study will be shared with manufacturers of investigational drugs, Ministry of Health, Labor and Welfare, and regulatory authorities related to pharmaceutical affairs.
  Data are attributed to Kyushu University and Daiichi Sankyo Co., Ltd. Protocols, informed consent form, and statistical analysis plans will be shared upon reasonable request.
  Contact: abe.kotaro.232@m.kyushu-u.ac.jp

REFERENCES:
- [Background] Hosokawa K, Abe K, Tsutsui H. Use of direct oral anticoagulants prevents increase in pulmonary vascular resistance and incidence of clinical worsening in patients with chronic thromboembolic pulmonary hypertension. Thromb Res. 2019 Aug;180:43-46. doi: 10.1016/j.thromres.2019.05.018. Epub 2019 May 31. No abstract available. PMID 31200342
- [Derived] Hosokawa K, Abe K, Kishimoto J, Kobayakawa Y, Todaka K, Tamura Y, Tatsumi K, Inami T, Ikeda N, Taniguchi Y, Minatsuki S, Murohara T, Yasuda S, Fukuda K, Tsutsui H. Efficacy and safety of edoxaban in patients with chronic thromboembolic pulmonary hypertension: protocol for a multicentre, randomised, warfarin-controlled, parallel group trial - KABUKI trial. BMJ Open. 2022 Jul 19;12(7):e061225. doi: 10.1136/bmjopen-2022-061225. PMID 37070473